CLINICAL TRIAL: NCT04255121
Title: Interest of the Alkalinization of the Adrenaline Lidocaine Solution for Conversion of Epidural Analgesia Into Epidural Anesthesia During an Emergency Caesarean
Brief Title: Bicarbonate Epidural Injection in Emergency Caesarian
Acronym: BiEpIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO19144*
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Emergency Caesarean
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alkalinization of adrenaline lidocaine solution arm (Experimental): conversion of epidural analgesia into epidural anesthesia during an emergency caesarean using an alkalinization of adrenaline lidocaine solution
  Interventions: Drug: 2% adrenaline lidocaine associated with 4.2% sodium bicarbonate
- adrenaline lidocaine solution arm (Active Comparator): conversion of epidural analgesia into epidural anesthesia during an emergency caesarean using a adrenaline lidocaine solution
  Interventions: Drug: 2% adrenaline lidocaine

INTERVENTIONS:
Drug: 2% adrenaline lidocaine associated with 4.2% sodium bicarbonate — conversion of epidural analgesia into epidural anesthesia during an emergency caesarean using an alkalinization of adrenaline lidocaine solution
  Arms: alkalinization of adrenaline lidocaine solution arm
Drug: 2% adrenaline lidocaine — conversion of epidural analgesia into epidural anesthesia during an emergency caesarean using an adrenaline lidocaine solution
  Arms: adrenaline lidocaine solution arm

SUMMARY:
During labor, pain is systematic. In France, epidural analgesia is the gold standard to fight pain.

Sometimes, emergency situations involve the maternal or fetal prognosis and require an emergency fetal extraction by caesarean. When an effective epidural analgesia is in place, an injection of adrenaline lidocaine converts this epidural analgesia into an epidural anesthesia allowing a surgical procedure. Sometimes, the time required to set up the anesthesia cannot be expected and a general anesthesia is performed.

Local anesthetics used during epidural analgesia have Pka between 7.8 and 8.1. In solution, local anesthetics exist in two forms: an un-ionized form and an ionized form. The non-ionized form is liposoluble and crosses the lipid membranes to reach the site of intracellular action. The non-ionized form conditions the time taken to install anesthesia.

When the pH of the solution is equal to Pka, un-ionized and ionized form are present in equal quantity. Commercial local anesthetic solutions have acidic pH and so contained a majority of ionized form. Alkalinization of local anesthetics solution should bring the pH closer to pKa and therefore to favor a greater proportion of non-ionized form.

DETAILED DESCRIPTION:
The aim of this study is to evaluate impact of an alkalinization of adrenaline lidocaine solution for conversion of epidural analgesia into epidural anesthesia during an emergency caesarean.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women followed up in the Reims University Hospital
* women whose birth is expected by vaginal delivery in the Reims University Hospital
* women wishing to benefit from epidural analgesia
* women agreeing to participate in the research and having signed informed consent
* women aged 18 years old and more
* women affiliated to a social security system

Exclusion Criteria:

* women who don't benefit from emergency caesarian (vaginal delivery or scheduled caesarian)
* women for whom epidural analgesia cannot be used
* women for whom epidural analgesia is not effective

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
delay in obtaining a T6 anesthetic level | 15 minutes
  delay to obtain a T6 anesthetic level evaluated in minute

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided